CLINICAL TRIAL: NCT01151553
Title: Comparative of Markers of Oxidative Stress Present Pre and Post Cardiac Resynchronization Therapy Outcome Predictors
Brief Title: Oxidative Stress Markers and Cardiac Resynchronization Therapy (CRT) Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding, lost support staff. No data collected/processed
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Heather Bloom, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012235
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Congestive Heart Failure
Keywords: Cardiology; Cardiomyopathy; Cardiovascular Disease; Cardiac Resynchronization Therapy (CRT)
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with CHF with CRT Therapy (Other): Patients with CHF with CRT Therapy
  Interventions: Device: CRT Therapy

INTERVENTIONS:
Device: CRT Therapy — Screen for enrollment criteria, consented, echocardiogram and electrocardiogram performed, demographics reviewed, obtain blood sample, pre-operative QOL questionnaire and 6 minute hall walk

SUMMARY:
This is a research study that is evaluating blood markers which may predict which patients who receive CRT will improve. Congestive heart failure (CHF) is associated with increased oxidative stress, a condition where abnormal oxygen forms are produced. These forms harm the cells of the heart and cause damage to the heart muscle. We would like to see if blood levels of these forms improve after CRT, and if they can be measured early after surgery to predict who will and who will not benefit from surgery.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a common diagnosis with significant clinical impact. Although medical therapy exists, many patients on optimal medical treatment are still highly symptomatic. About 1/3 of these patients have a condition known as "dyssynchrony", where the walls of the heart beat in an uncoordinated way, causing worsening of CHF symptoms. A newer therapy known as cardiac resynchronization therapy (CRT) has been successful in decreasing symptoms in these dyssynchronous patients. It involves surgical placement of a pacemaker containing 3 wires- one in the top part of the heart (atrium) to coordinate the top and bottom parts of the heart beat, and two on the bottom to coordinate the bottom parts of the heart beat (ventricles). This treatment, however, does not work for up to 1/3 of patients with dyssynchrony.

Recent studies have found that CHF is associated with increased oxidative stress. This is a condition where abnormal oxygen forms are produced. These forms harm the cells of the heart, causing them to beat abnormally and causing damage to the heart muscle. We would like to see if levels of these forms improve after CRT, and if they can be measured early after surgery to predict who will and who will not benefit from surgery.

In this study, we will compare blood markers of oxidative stress between patients with CHF and an already-collected set of control patients to confirm these levels are elevated at baseline. Then, we will perform CRT surgery and implant pacemakers in the CHF patients. At 1 week and 3 months postoperatively, we will measure blood markers again, and see if they have improved in patients whose symptoms have improved. Patients will undergo echocardiograms to document their abnormal hearts, do a 6 minute hall walk to measure their exercise tolerance, and take a standardized questionnaire to measure their symptoms of CHF. These test results will be compared pre and post CRT to assess response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Screen for enrollment criteria,
* Consented,
* Echocardiogram and electrocardiogram performed,
* Demographics reviewed,
* Obtain blood sample,
* Pre-operative QOL questionnaire.

Exclusion Criteria:

* 6 minute hall walk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Bloom, MD, FACC, Principal Investigator — Emory University IRB

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With CHF With CRT Therapy: Patients with CHF with CRT Therapy
  CRT Therapy : Screen for enrollment criteria, consented, echocardiogram and electrocardiogram performed, demographics reviewed, obtain blood sample, pre-operative QOL questionnaire and 6 minute hall walk
Period: Overall Study
Arm/Group | Patients With CHF With CRT Therapy
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With CHF With CRT Therapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Markers of Oxidative Stress Pre and Post Cardiac Resynchronization Therapy as Outcome
Description: Patient has a weak heart and scheduled to have CRT placed in the next month. The study is to evaluate blood markers which may predict which patients who receive CRT will improve
Time Frame: One year
Population: Early termination leading to small numbers of subjects; lost funding and staff, no data collected/processed.
Arm/Group | Patients With CHF With CRT Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: "0" Total Number of Participants at Risk reported since serious and/or other [non-serious] adverse events were not collected/assessed.
Arm/Group | Patients With CHF With CRT Therapy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects; lost funding and staff, no data collected/processed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No